CLINICAL TRIAL: NCT01546259
Title: Water Method With Water Exchange Versus Air Insufflation in Low-BMI Female Patients Undergoing Unsedated Colonoscopy: a Prospective Randomized, Controlled Trial
Brief Title: Water Method in Low-body Mass Index (BMI) Female Patients With Unsedated Colonoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 20120216-7
Record Dates: First submitted 2012-02-24; First posted 2012-03-07 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Adenoma; Pain
Keywords: colonoscopy; water; female; BMI; unsedated; low BMI female patients; Intubation
MeSH Terms: conditions — Adenoma; Pain | interventions — Water; Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air colonoscopy (No Intervention): Colonoscopy will be performed without medications and with judicious air insufflation during colonoscope insertion.
- Water colonoscopy (Other): Colonoscopy will be performed without medications and aided by water infusion in-lieu of air insufflation during insertion of the colonoscope.
  Interventions: Other: Water colonoscopy

INTERVENTIONS:
Other: Water colonoscopy — Colonoscopy will be performed without medications and aided by water infusion in-lieu of air insufflation during insertion of the colonoscope. The water infusion involves putting warm sterile water into the colon to open up the colon for advancement of the colonoscope until the end of the colon (cecum) is reached. The water is delivered through scope irrigation channel by an infusion pump equipped with a foot switch which will be controlled by the endoscopist. Infused water used to cleanse residual fecal matter will be suctioned as needed to clear the colonic lumen.
  Other Names: Water; colonoscopy
  Arms: Water colonoscopy

SUMMARY:
Water method with water exchange has been shown to reduce medication requirement and pain experienced during colonoscopy. It increases the success rate of cecal intubation in sedated and unsedated patients undergoing screening colonoscopy. Exchange of water during scope insertion minimizes distension of the colonic lumen and decreases loop formation. Exclusion of air from the colon during insertion by omission of air insufflations and suction removal of residual air prevent elongation of the colon. These maneuvers facilitate colonoscopy insertion in average patients and may enhance the success of difficult colonoscopy.

Female gender and low-body mass index (BMI) is independently associated with incomplete colonoscopy, respectively. The investigators postulate that low-BMI female patients may benefit from using the water method for colonoscopy. In this proposal the investigators test the hypothesis that compared with conventional air insufflations the water method with water exchange significantly enhances the success rate of cecal intubation in low-BMI female patients.

The aim of the study is to compare the outcome of colonoscopy using the water method versus the conventional air method in low-BMI female patients. The primary outcome is cecal intubation success rate. The secondary outcomes include cecal intubation time, maximum pain score during colonoscopy, overall pain score after colonoscopy and adenoma detection rate.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with BMI < 20

Exclusion Criteria:

* History of colorectal surgery
* Severe colonic stricture or obstructing tumor
* Patients who cannot give informed consent and those who are hemodynamically unstable

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Cecal intubation success rate | up to two years
  Insertion of a colonoscope to the cecum

SECONDARY OUTCOMES:
Adenoma detection rate | up to two years
  The proportion of participants with at least one adenoma in each group
Pain Scores on the Visual Analog Scale | up to two years
  0 = no pain, to 10 = most severe pain
Cecum intubation time | up to two years
  Total time of colonoscope intubation from anus to cecum

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, MD, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China